CLINICAL TRIAL: NCT01252342
Title: Does Intramyometrial Oxytocin Improve Outcome in Elective Cesarean Delivery?
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Proposed doses were too large, bolus oxytocin may cause cases of arrythmias, and some even advocate slowing down the infusion rates that are currently used.
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Oxytocin
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-10

CONDITIONS: Postpartum Hemorrhage; Uterine Atony
Keywords: Oxytocin; Intramyometrial
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Intramyometrial oxytocin (Experimental)
  Interventions: Drug: Oxytocin
- Intramyometrial Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — 10 U intramyometrial oxytocin bolus immediately after cesarian delivery, and an infusion of 20 U/L of oxytocin at 500ml/hr.
  Arms: Intramyometrial oxytocin
Drug: Saline — 10U intramyometrial normal saline bolus immediately after cesarian delivery, and an infusion of 20U/L of oxytocin at 500ml/hr.
  Arms: Intramyometrial Saline

SUMMARY:
Oxytocin use has become routine practice in elective cesarean delivery to promote uterine contraction and reduce blood loss. However, there is a lack of consensus regarding the best dose of oxytocin and the most effective route of administration. Most dosage and delivery systems have been empirically derived.

It is currently our practice at the Royal University Hospital to start an oxytocin infusion (20U/L) once the baby has been delivered. Some anesthesiologists use bolus intravenous oxytocin and it is occasionally requested by the obstetrician. A few obstetricians also choose to inject bolus oxytocin directly into the uterus (intramyometrial).

The primary objectives of the study include:

1. Determine if our standard 'low dose' oxytocin infusion is adequate prophylaxis to prevent need for additional uterotonics, including additional oxytocin;
2. Determine if the addition of prophylactic intramyometrial oxytocin improves both the primary outcome (uterine tone) and secondary outcomes (estimated blood loss, preoperative to postoperative change in hematocrit, need for additional uterotonics, and need for blood pressure support); and
3. Act as a dose finding study to determine if the intramyometrial dose is sufficient to augment uterine contraction.

The working hypothesis is that the use of intramyometrial oxytocin will not improve primary or secondary outcomes compared to the current practice of an oxytocin infusion alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Parturients
* Elective cesarean Delivery
* Term (> 37 wks gestational age) as defined by ultrasound or last menstrual period
* Singleton fetus
* Vertex presentation
* Age > 18
* BMI < 40
* Height > 5'2" and < 5"8"
* Written informed consent

Exclusion Criteria:

* Placenta previa
* Multiple gestation
* Preeclampsia
* Gestational Diabetes or pre-existing diabetes
* Macrosomia (estimated fetal weight prior to delivery)
* Polyhydramnios
* Oligohydramnios
* Uterine fibroids
* More than 2 previous cesarean deliveries
* Suspected adherent placenta (acreta/increta/percreta)
* Planned general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Uterine Tone | The blinded obstetrician will assess uterine tone at 1,2,4,6, 8 and 10-minute intervals

SECONDARY OUTCOMES:
Estimated Blood Loss | Immediately Post-operatively
Pre-operative to post-operative change in hematocrit | 24 hrs post-operative
Need for additional unterotonics | Immediately post delivery
Need for blood pressure support | Intra-operative period following administration of oxytocin

CONTACTS AND LOCATIONS:
Overall Officials: Monica K San Vicente, MD, Study Director — University of Saskatchewan, Department of Anesthesia; David C Campbell, MD, FRCPC, Principal Investigator — University of Saskatchewan, Department of Anesthesia
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada